CLINICAL TRIAL: NCT02810119
Title: A Randomized, Double-Blind, Placebo-Controlled, Pilot Study to Evaluate the Efficacy and Safety of LO2A Eye Drops in Patients With Moderate to Severe Conjunctivochalasis
Brief Title: To Evaluate the Efficacy and Safety of LO2A Eye Drops in Patients With Conjunctivochalasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuwize LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WP-LO2A-02
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Conjunctivochalasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LO2A (Experimental): Sodium Hyaluronate
  Interventions: Drug: LO2A
- Placebo-Controlled Saline (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LO2A
  Arms: LO2A
Drug: Placebo
  Arms: Placebo-Controlled Saline

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Pilot Study to Evaluate the Efficacy and Safety of LO2A Eye Drops in Patients with Moderate to Severe Conjunctivochalasis

DETAILED DESCRIPTION:
Phase 2a, randomized, placebo-controlled, pilot study in up to 21 adult patients with moderate to severe CCh. Eligible patients will be randomly assigned in a 2:1 (active:placebo) ratio to one of two treatment groups, LO2A or placebo.

This study with 4 visits, will consist of a screening period of up to 2 weeks and a 3-month treatment period (topical, OU, QID application of eye drops).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race and ≥ 18 years of age.
2. Willing and able to provide voluntary written informed consent.
3. Moderate to severe conjunctivochalasis defined by:

   * LIPCOF score ≥ 2; and
   * Lissamine green conjunctival staining score ≥ 5 according to National Eye Institute/Industry Workshop report.
4. Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Subject has concurrent, uncontrolled medical condition, or psychiatric illness which could place him/her at unacceptable risk, including, but not limited to:

   * Subject has been diagnosed or treated for another malignancy within 3 years of screening, except in situ malignancy, or low-risk prostate, skin or cervix cancer after curative therapy.
   * A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications.
2. Subjects with pterygium.
3. Subjects with active, allergic keratoconjunctivitis, or conjunctivitis of infectious origin.
4. Subjects with blepharitis requiring treatment.
5. Subjects with a history of surgery affecting the eye surface, as well as eye injuries within 3 months of screening.
6. Subjects currently using any topical ophthalmic treatment (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial.
7. Subjects who have used any of the following medications or treatments:

   * LASIK or PRK surgery within 12 months of Visit 1.
   * Use of contact lenses within 7 days of Visit 1.
   * Punctal plug insertion within 30 days of Visit 1.
   * Use of topical or systemic cyclosporine within 30 days of Visit 1.
   * Use of medications known to cause ocular drying (e.g. antihistamines, sleep aids, etc.), unless at a stable dose, within 30 days of Visit 1.
8. Known hypersensitivity to sodium hyaluronate or any LO2A excipients (glycerol and Carbomer 981).
9. Active abuse of alcohol or drugs.
10. Any condition, which in the opinion of the Investigator, would place the patient at an unacceptable risk if participating in the study protocol.
11. Participation in a clinical trial of an investigational (unapproved) drug or device within 1 month prior to screening or scheduled to receive another investigational drug or device during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in lissamine green conjunctival staining (LGCS) score | baseline and 3 months

SECONDARY OUTCOMES:
The change in the lid-parallel conjunctival fold (LIPCOF) grade score at 1 and 3 months compared to baseline | baseline, 1 month and 3 months
The change from baseline in LGCS score | baseline and 1 month
The change in tear-film break up time (TFBUT) compared to baseline at 1 and 3 months | baseline, 1 month and 3 months]
The change in ocular surface disease index (OSDI) questionnaire score compared to baseline at 1 and 3 months | baseline, 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai MC, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Final Data report will be publish when the study will be finalized